CLINICAL TRIAL: NCT02949804
Title: Relation Between Vasovagal Tendency and Smoking Among University Students
Status: Completed | Type: Observational
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Sponsor
Other Study IDs: 2
Record Dates: First submitted 2016-10-26; First posted 2016-10-31 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Vasovagal Syncope; Smoke Inhalation
MeSH Terms: conditions — Syncope, Vasovagal; Smoke Inhalation Injury

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Smoker: Vasovagal tendency will be compared among smokers and non smokers
  Interventions: Behavioral: Comparison between two groups
- Non-smokers: Vasovagal tendency will be compared among smokers and non smokers
  Interventions: Behavioral: Comparison between two groups

INTERVENTIONS:
Behavioral: Comparison between two groups — Comparison will be made between smokers and non smokers regarding vasovagal tendency

SUMMARY:
Almost everyone is aware these days is aware about the risk of smoking. Still many people start this habit specially in early life and during college year. We aim to investigate in this study if there is a drive to smoke in people with vasovagal tendency to improve their symptoms, even if not aware of this. Vasovoagal symptoms are common and include dizziness, smoking, sweating, abdominal pain, fatigue and syncope. Some studies have shown correlation between smoking and a positive tilt table test which is indicative of vasovagal tendency. By collecting the information regarding smoking habit and vasovagal symptoms analysis can be done to see if there is correlation between these two factors

DETAILED DESCRIPTION:
Methods

A questionnaire will be conducted among university students to investigate the tendency toward vasovagal symptoms and also smoking habits. Statistical correlation will be subsequently conducted to see if there is correlation between those two problems (vasovagal symptoms and smoking)

Study criteria inclusion

Benefit to the patient:

There is no direct benefit for participation in the study. The information obtained may help in the future to find factors that increase smoking and being aware of these factors may help in controlling the habit of smoking.

ELIGIBILITY:
Inclusion Criteria:

* College students who agree to participate in the questionnaire

Exclusion Criteria:

* Unable or does not consent to fill the form

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Students at the university or college
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-12; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Incidence of vasovagal tenancy in smokers and non smokers | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Munir Al Zaqqa, MD, Principal Investigator — Jordan Collaborating Cardiology Group
Locations (1):
- Istishari hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
Once data is collected it will be shared with researchers after making individuals anonymous